CLINICAL TRIAL: NCT04177355
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of HIV-1 BG505 SOSIP.664 gp140 With TLR Agonist and/or Aalum Adjuvants and VRC HIV Env Trimer 4571 and 3M-052-AF With Alum in Healthy, HIV-uninfected Adults
Brief Title: Evaluating the Safety and Immunogenicity of HIV-1 BG505 SOSIP.664 gp140 With TLR Agonist and/or Alum Adjuvants in Healthy, HIV-uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); International AIDS Vaccine Initiative (Network); Access to Advanced Health Institute (AAHI) (Other); Dynavax Technologies Corporation (Industry); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 137; 38559 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — 1018 oligonucleotide; aluminum sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Part A, Group 1 (T1): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum (Experimental): Participants will receive 100 mcg of BG505 SOSIP.664 gp140, admixed with 1 mcg of 3M-052-AF and 500 mcg of Aluminum Hydroxide Suspension (Alum), as one intramuscular (IM) injection at Months 0 and 2, with optional second boost at Month 6.
  Interventions: Biological: BG505 SOSIP.664 gp140; Biological: 3M-052-AF; Biological: Alum (Aluminum Hydroxide Suspension)
- Part A, Group 1 (P1): Placebo (Placebo Comparator): Participants will receive placebo as one IM injection at Months 0 and 2, with optional second boost at Month 6.
  Interventions: Biological: Placebo
- Part A, Group 2 (T2): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum (Experimental): Participants will receive 100 mcg of BG505 SOSIP.664 gp140, admixed with 5 mcg of 3M-052-AF and 500 mcg of Alum, as one IM injection at Months 0 and 2, with optional second boost at Month 6.
  Interventions: Biological: BG505 SOSIP.664 gp140; Biological: 3M-052-AF; Biological: Alum (Aluminum Hydroxide Suspension)
- Part A, Group 2 (P2): Placebo (Placebo Comparator): Participants will receive placebo as one IM injection at Months 0 and 2, with optional second boost at Month 6.
  Interventions: Biological: Placebo
- Part B, Group 3 (T3): BG505 SOSIP.664 gp140 + CpG 1018 + Alum (Experimental): Participants will receive 100 mcg of BG505 SOSIP.664 gp140, admixed with 300 mcg of CpG 1018 and 500 mcg of Alum, as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: BG505 SOSIP.664 gp140; Biological: CpG 1018; Biological: Alum (Aluminum Hydroxide Suspension)
- Part B, Group 3 (P3): Placebo (Placebo Comparator): Participants will receive placebo as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: Placebo
- Part B, Group 4 (T4): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum (Experimental): Participants will receive 100 mcg of BG505 SOSIP.664 gp140, admixed with either 1 mcg or 5 mcg of 3M-052-AF (the highest tolerated dose from Part A), and 500 mcg of Alum, as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: BG505 SOSIP.664 gp140; Biological: 3M-052-AF; Biological: Alum (Aluminum Hydroxide Suspension)
- Group 4 (P4): Placebo (Placebo Comparator): Participants will receive placebo as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: Placebo
- Part B, Group 5 (T5): BG505 SOSIP.664 gp140 + GLA-LSQ (Experimental): Participants will receive 100 mcg of BG505 SOSIP.664 gp140, admixed with GLA-LSQ (GLA 5 mcg, and QS-21 2 mcg), as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: BG505 SOSIP.664 gp140; Biological: GLA-LSQ
- Part B, Group 5 (P5): Placebo (Placebo Comparator): Participants will receive placebo as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: Placebo
- Part B, Group 6 (T6): BG505 SOSIP.664 gp140 + Alum (Experimental): Participants will receive 100 mcg of BG505 SOSIP.664 gp140, admixed with 500 mcg of Alum, administered as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: BG505 SOSIP.664 gp140; Biological: Alum (Aluminum Hydroxide Suspension)
- Part B, Group 6 (P6): Placebo (Placebo Comparator): Participants will receive placebo as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: Placebo
- Part C, Group 7 (T7): BG505 SOSIP.664 gp140 + Alum (Experimental): Participants will receive BG505 SOSIP.664 gp140, 100 mcg admixed with 3M-052-AF, 3 mcg and Alum, 500 mcg to be administered as one 0.5-mL dose intramuscularly (IM) at months 0, 2, and 6.
  Interventions: Biological: BG505 SOSIP.664 gp140; Biological: 3M-052-AF; Biological: Alum (Aluminum Hydroxide Suspension)
- Part C, Group 7 (P7): Placebo (Placebo Comparator): Participants will receive placebo as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: Placebo
- Part C, Group 8 (T8): Trimer 4571 + Alum (Experimental): Participants will receive Trimer 4571, 100 mcg admixed with 3M-052-AF, 5 mcg and Alum, 500 mcg to be administered as one 0.5-mL dose IM at months 0, 2, and 6.
  Interventions: Biological: 3M-052-AF; Biological: Alum (Aluminum Hydroxide Suspension); Biological: Trimer 4571
- Part C, Group 8 (P8): Placebo (Placebo Comparator): Participants will receive placebo as one IM injection at Months 0, 2, and 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BG505 SOSIP.664 gp140 — Administered by IM injection
  Arms: Part A, Group 1 (T1): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part A, Group 2 (T2): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part B, Group 3 (T3): BG505 SOSIP.664 gp140 + CpG 1018 + Alum; Part B, Group 4 (T4): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part B, Group 5 (T5): BG505 SOSIP.664 gp140 + GLA-LSQ; Part B, Group 6 (T6): BG505 SOSIP.664 gp140 + Alum; Part C, Group 7 (T7): BG505 SOSIP.664 gp140 + Alum
Biological: Placebo — Administered by IM injection
  Arms: Group 4 (P4): Placebo; Part A, Group 1 (P1): Placebo; Part A, Group 2 (P2): Placebo; Part B, Group 3 (P3): Placebo; Part B, Group 5 (P5): Placebo; Part B, Group 6 (P6): Placebo; Part C, Group 7 (P7): Placebo; Part C, Group 8 (P8): Placebo
Biological: 3M-052-AF — Administered by IM injection
  Arms: Part A, Group 1 (T1): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part A, Group 2 (T2): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part B, Group 4 (T4): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part C, Group 7 (T7): BG505 SOSIP.664 gp140 + Alum; Part C, Group 8 (T8): Trimer 4571 + Alum
Biological: CpG 1018 — Administered by IM injection
  Arms: Part B, Group 3 (T3): BG505 SOSIP.664 gp140 + CpG 1018 + Alum
Biological: GLA-LSQ — Administered by IM injection
  Arms: Part B, Group 5 (T5): BG505 SOSIP.664 gp140 + GLA-LSQ
Biological: Alum (Aluminum Hydroxide Suspension) — Administered by IM injection
  Arms: Part A, Group 1 (T1): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part A, Group 2 (T2): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part B, Group 3 (T3): BG505 SOSIP.664 gp140 + CpG 1018 + Alum; Part B, Group 4 (T4): BG505 SOSIP.664 gp140 + 3M-052-AF + Alum; Part B, Group 6 (T6): BG505 SOSIP.664 gp140 + Alum; Part C, Group 7 (T7): BG505 SOSIP.664 gp140 + Alum; Part C, Group 8 (T8): Trimer 4571 + Alum
Biological: Trimer 4571 — Administered by IM injection
  Arms: Part C, Group 8 (T8): Trimer 4571 + Alum

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of HIV-1 BG505 SOSIP.664 gp140 with TLR agonist and/or alum adjuvants in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of HIV-1 BG505 SOSIP.664 gp140 with TLR agonist and/or alum adjuvants in healthy, HIV-uninfected adults.

The study will be conducted in three parts (Part A, B and C). Part A will include two groups (Groups 1 and 2), Part B will include four groups (Groups 3, 4, 5, and 6) and Part C will include two groups (Groups 7 and 8).

Participants in Part A will be randomly assigned to receive the BG505 SOSIP.664 gp140 vaccine admixed with 3M-052-AF and alum adjuvant or to receive placebo. Part A participants will be enrolled sequentially in Groups 1 and 2 for dose escalation.

Participants in Part B will be randomly assigned to Groups 3, 4, 5, or 6, to receive the BG505 SOSIP.664 gp140 vaccine with an adjuvant (the specific adjuvant will vary by group) or to receive placebo.

Participants in Part C will be randomly assigned to Groups 7 or 8 to receive:

Group 7: The same BG505 SOSIP immunogen but with a lower dose (3mcg) of 3M-052-AF + Alum, Group 8: The Trimer 4571 with 5mcg 3M-052-AF + Alum, or to receive placebo.

Participants in Part A will attend 8 months of scheduled clinic visits, and they will be contacted by study staff at Month 14 for follow-up health monitoring. Upon protocol amendment, subjects in Part A were invited to receive a third immunization.

Participants in Part B will attend 18 months of scheduled clinic visits. Participants in Part C will attend 18 months of scheduled clinic visits.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 through 50 years, inclusive
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent until after the final study contact.
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit (see study protocol for more information)

Laboratory Inclusion Values

Hemogram/Complete blood count (CBC)

* Hemoglobin

  * ≥ 11.0 g/dL for volunteers who were assigned female sex at birth
  * ≥ 13.0 g/dL for volunteers who were assigned male sex at birth and transgender males who have been on hormone therapy for more than 6 consecutive months
  * ≥ 12.0 g/dL for transgender females who have been on hormone therapy for more than 6 consecutive months
  * For transgender volunteers who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on the sex assigned at birth.
* White blood cell count = 2,500 to 12,000 cells/mm^3 with normal differential, or differential approved by Investigator of Record (IoR) or designee as not clinically significant
* Total lymphocyte count ≥ 650 cells/mm^3 with normal differential, or differential approved by IoR or designee as not clinically significant
* Remaining differential either within institutional normal range or with IoR or designee approval
* Platelets = 125,000 to 550,000 cells/mm^3

Chemistry

* Alanine aminotransferase (ALT) < 1.25 times the institutional upper limit of normal
* Creatinine < 1.1 times the institutional upper limit of normal

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative U.S. Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (If trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range,)

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test at screening (ie, prior to randomization) and prior to study product administration or any optional study procedure (eg, leukapheresis, fine needle aspirate, bone marrow aspiration, mucosal secretion collection or mucosal biopsy) on the day of study product administration or procedure. Persons who are NOT of reproductive potential due to having undergone hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was assigned female sex at birth:

  * Must agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until 6 months after the final study vaccination. Effective contraception is defined as using the following methods:

    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,
    * Intrauterine device (IUD),
    * Hormonal contraception,
    * Tubal ligation, or
    * Any other contraceptive method approved by the HVTN 137 Protocol Safety Review Team (PSRT)
    * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy or bilateral oophorectomy;
  * Or be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until 6 months after the last vaccination.

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) ≥ 40; or BMI ≥ 35 with 2 or more of the following: age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 137 study
* Pregnant or breastfeeding
* Active duty and reserve US military personnel

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 137 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational; the HVTN 137 PSRT will determine eligibility on a case-by-case basis
* Non-HIV experimental vaccine(s) received within the last 1 year in a prior vaccine trial. Exceptions may be made by the HVTN 137 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 137 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 1 year ago, eligibility for enrollment will be determined by the HVTN 137 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first vaccination or scheduled within 30 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination or scheduled for 14 days after injection (eg, tetanus, pneumococcal, hepatitis virus A or B)
* Previous receipt of HEPLISAV, Shingrix, or RTS,S/AS01B/Mosquirix vaccine received within 30 days prior to first vaccination or scheduled for 30 days after injection.
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses ≤ 60 mg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment)
* Serious adverse reactions to vaccines or to vaccine components, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a non-anaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination (for mAb see criterion above)
* Autoimmune disease, current or history
* AESIs: Volunteers who currently have, or have a history of, any condition that could be considered an AESI for the product(s) administered in this protocol (representative examples are listed in the study protocol)
* Immunodeficiency

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:

    * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma
* Diabetes mellitus type 1 or type 2 (Not exclusionary: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined in this protocol as consistently < 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
* Bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of generalized urticaria, angioedema, or anaphylaxis. (Not exclusionary: angioedema or anaphylaxis to a known trigger with at least 5 years since last reaction to demonstrate satisfactory avoidance of trigger.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Juliana McElrath, Study Chair — Seattle Vaccine Trials Unit; Nadine Rouphael, Study Chair — Emory University
Locations (10):
- United States (10):
  - Alabama CRS, Birmingham, Alabama
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS (Site 31801), New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahn WO, Parks KR, Shen M, Ozorowski G, Janes H, Ballweber-Fleming L, Woodward Davis AS, Duplessis C, Tomai M, Dey AK, Sagawa ZK, De Rosa SC, Seese A, Kallur Siddaramaiah L, Stamatatos L, Lee WH, Sewall LM, Karlinsey D, Turner HL, Rubin V, Furth S, MacPhee K, Duff M, Corey L, Keefer MC, Edupuganti S, Frank I, Maenza J, Baden LR, Hyrien O, Sanders RW, Moore JP, Ward AB, Tomaras GD, Montefiori DC, Rouphael N, McElrath MJ. Use of 3M-052-AF with Alum adjuvant in HIV trimer vaccine induces human autologous neutralizing antibodies. J Exp Med. 2024 Oct 7;221(10):e20240604. doi: 10.1084/jem.20240604. Epub 2024 Sep 5. PMID 39235529

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Group T1: BG505 SOSIP.664 gp140 & (1 mcg 3M-052-AF + Alum) mo(0,2)
- Part A, Group T2: BG505 SOSIP.664 gp140 & (5 mcg 3M-052-AF + Alum) mo(0,2)
- Part A, Group C1: Placebo for BG505 SOSIP.664 gp140 & adjuvant mo(0,2)
- Part B, Group T3: BG505 SOSIP.664 gp140 & (CpG 1018 + Alum) mo(0,2,6)
- Part B, Group T4: BG505 SOSIP.664 gp140 & (3M-052-AF + Alum) mo(0,2,6)
- Part B, Group T5: BG505 SOSIP.664 gp140 & GLA-LSQ mo(0,2,6)
- Part B, Group T6: BG505 SOSIP.664 gp140 & Alum mo(0,2,6)
- Part B, Group C2: Placebo for BG505 SOSIP.664 gp140 & adjuvant mo(0,2,6)
- Part B, Group T7: BG505 SOSIP.664 gp140 & (3mcg 3M-052-AF+Alum) mo(0,2,6)
- Part B, Group T8: Trimer 4571 & (5mcg 3M-052-AF+Alum) mo(0,2,6)
- Part B, Group C3: Placebo for BG505 SOSIP.664 gp140/Trimer 4571 & adjuvant mo(0,2,6)
Period: Overall Study
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part B, Group T7 | Part B, Group T8 | Part B, Group C3
Started | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Safety Population | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Received Optional Second Boost at 6 Months (Part A) | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 5 | 8 | 2 | 18 | 16 | 20 | 19 | 9 | 9 | 10 | 2
Not Completed | 0 | 2 | 0 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part C, Group T7: BG505 SOSIP.664 gp140 & (3mcg 3M-052-AF+Alum) mo(0,2,6)
- Part C, Group T8: Trimer 4571 & (5mcg 3M-052-AF+Alum) mo(0,2,6)
- Part C, Group C3: Placebo for BG505 SOSIP.664 gp140/Trimer 4571 & adjuvant mo(0,2,6)
- Total: Total of all reporting groups
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part C, Group T7 | Part C, Group T8 | Part C, Group C3 | Total
Number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2 | 127
Age, Continuous [Median (Full Range); unit: years] | 28 [21 to 35] | 25.5 [20 to 34] | 23.5 [23 to 24] | 28 [21 to 43] | 32 [19 to 50] | 28 [18 to 48] | 26.5 [20 to 48] | 33 [19 to 49] | 30 [23 to 48] | 36 [27 to 46] | 44 [41 to 47] | 29 [18 to 50]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-20 years | 0 | 1 | 0 | 0 | 2 | 3 | 2 | 1 | 0 | 0 | 0 | 9
  21-30 years | 4 | 7 | 2 | 12 | 7 | 10 | 10 | 3 | 5 | 4 | 0 | 64
  31-40 years | 1 | 2 | 0 | 7 | 6 | 4 | 4 | 3 | 4 | 5 | 0 | 36
  41-50 years | 0 | 0 | 0 | 1 | 4 | 3 | 4 | 2 | 1 | 1 | 2 | 18
  Above 50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 2 | 13 | 9 | 12 | 8 | 3 | 7 | 6 | 1 | 71
  Male | 1 | 4 | 0 | 7 | 10 | 8 | 12 | 6 | 3 | 4 | 1 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 3 | 2 | 3 | 0 | 1 | 1 | 0 | 13
  Not Hispanic or Latino | 5 | 9 | 1 | 19 | 16 | 18 | 17 | 9 | 9 | 9 | 2 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 3 | 0 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 2 | 5 | 1 | 16
  White | 3 | 8 | 1 | 16 | 12 | 18 | 16 | 9 | 5 | 5 | 0 | 93
  More than one race | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2 | 127

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Solicited Adverse Events Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured for 7 days after each injection in Parts A and B and 14 days after each injection in Part C, up to Month 6
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part C, Group T7 | Part C, Group T8 | Part C, Group C3
Number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Participants
  None | 0 | 0 | 1 | 5 | 0 | 4 | 1 | 4 | 0 | 0 | 2
  Mild | 4 | 4 | 1 | 14 | 12 | 15 | 19 | 5 | 6 | 6 | 0
  Moderate | 1 | 6 | 0 | 1 | 7 | 1 | 0 | 0 | 4 | 4 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Solicited Adverse Events Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured for 7 days after each injection in Parts A and B and 14 days after each injection in Part C, up to Month 6
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part C, Group T7 | Part C, Group T8 | Part C, Group C3
Number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Participants
  Erythema/Redness: None | 5 | 8 | 2 | 19 | 19 | 20 | 20 | 9 | 9 | 10 | 2
  Erythema/Redness: Mild | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Erythema/Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: Severe | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: None | 4 | 8 | 2 | 20 | 16 | 20 | 19 | 9 | 9 | 9 | 2
  Induration/Swelling: Mild | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Induration/Swelling: Moderate | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Severe | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 4 | 8 | 2 | 19 | 16 | 20 | 19 | 9 | 9 | 9 | 2
  Erythema and/or Induration: Mild | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Erythema and/or Induration: Moderate | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Severe | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Solicited Adverse Events Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured for 7 days after each injection in Parts A and B and 14 days after each injection in Part C, up to Month 6
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part C, Group T7 | Part C, Group T8 | Part C, Group C3
Number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Participants
  Malaise and/or fatigue: None | 0 | 0 | 2 | 6 | 1 | 5 | 7 | 3 | 1 | 0 | 1
  Malaise and/or fatigue: Mild | 2 | 2 | 0 | 11 | 9 | 11 | 9 | 6 | 2 | 2 | 1
  Malaise and/or fatigue: Moderate | 2 | 5 | 0 | 3 | 5 | 4 | 4 | 0 | 6 | 7 | 0
  Malaise and/or fatigue: Severe | 1 | 3 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 1 | 1 | 2 | 16 | 2 | 13 | 15 | 6 | 1 | 2 | 2
  Myalgia: Mild | 1 | 2 | 0 | 4 | 5 | 4 | 5 | 3 | 4 | 2 | 0
  Myalgia: Moderate | 2 | 6 | 0 | 0 | 10 | 3 | 0 | 0 | 5 | 5 | 0
  Myalgia: Severe | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 0 | 0 | 2 | 10 | 2 | 12 | 10 | 5 | 2 | 1 | 2
  Headache: Mild | 3 | 4 | 0 | 10 | 12 | 5 | 7 | 4 | 4 | 3 | 0
  Headache: Moderate | 2 | 5 | 0 | 0 | 5 | 3 | 3 | 0 | 3 | 5 | 0
  Headache: Severe | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 3 | 3 | 2 | 17 | 7 | 16 | 15 | 9 | 3 | 2 | 2
  Nausea: Mild | 2 | 5 | 0 | 2 | 9 | 2 | 5 | 0 | 5 | 4 | 0
  Nausea: Moderate | 0 | 2 | 0 | 1 | 3 | 2 | 0 | 0 | 2 | 4 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 2 | 4 | 2 | 17 | 3 | 14 | 19 | 8 | 0 | 5 | 2
  Chills: Mild | 1 | 1 | 0 | 3 | 8 | 6 | 1 | 1 | 6 | 2 | 0
  Chills: Moderate | 1 | 5 | 0 | 0 | 6 | 0 | 0 | 0 | 4 | 2 | 0
  Chills: Severe | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 2 | 3 | 2 | 20 | 5 | 17 | 16 | 9 | 2 | 5 | 2
  Arthralgia: Mild | 1 | 4 | 0 | 0 | 6 | 3 | 4 | 0 | 5 | 3 | 0
  Arthralgia: Moderate | 1 | 3 | 0 | 0 | 7 | 0 | 0 | 0 | 3 | 1 | 0
  Arthralgia: Severe | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 0 | 0 | 2 | 6 | 1 | 4 | 4 | 2 | 0 | 0 | 1
  Max. Systemic Symptoms: Mild | 1 | 2 | 0 | 10 | 4 | 10 | 10 | 7 | 3 | 1 | 1
  Max. Systemic Symptoms: Moderate | 3 | 5 | 0 | 4 | 9 | 6 | 6 | 0 | 5 | 8 | 0
  Max. Systemic Symptoms: Severe | 1 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 2 | 1 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 3 | 6 | 2 | 18 | 3 | 20 | 20 | 9 | 8 | 7 | 2
  Temperature: Mild | 2 | 1 | 0 | 2 | 11 | 0 | 0 | 0 | 2 | 2 | 0
  Temperature: Moderate | 0 | 3 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Local Laboratory Values Meeting Grade 1 AE Criteria or Above
Description: For each local laboratory measure meeting Grade 1 AE criteria (Mild) or above as specified in the DAIDS AE Grading Table, counts of severity were presented by treatment group and timepoint for the overall population
Time Frame: Measured through Month 8 (Part A without second boost) or Month 12 (Part A with second boost, Part B, Part C)
Population: Overall Number of Participants Analyzed represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part C, Group T7 | Part C, Group T8 | Part C, Group C3
Number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Participants
  Neutrophils (1000 cells/cubic mm)- Day 14: number analyzed (Participants) | 5 | 10 | 2 | 20 | 18 | 20 | 20 | 9 | 10 | 10 | 2
  Neutrophils (1000 cells/cubic mm)- Day 14 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (g/dL)- Day 182 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
  Hemoglobin (g/dL)- Day 364: number analyzed (Participants) | 5 | 10 | 2 | 19 | 19 | 20 | 20 | 9 | 10 | 10 | 2
  Hemoglobin (g/dL)- Day 364 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 14: number analyzed (Participants) | 5 | 8 | 2 | 20 | 19 | 20 | 19 | 9 | 10 | 10 | 2
  ALT (SGPT) (U/L)- Day 14 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 70: number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 6 | 10 | 10 | 2
  ALT (SGPT) (U/L)- Day 70 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 182: number analyzed (Participants) | 3 | 10 | 2 | 20 | 19 | 20 | 20 | 8 | 10 | 10 | 2
  ALT (SGPT) (U/L)- Day 182 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  ALT (SGPT) (U/L)- Day 364: number analyzed (Participants) | 3 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
  ALT (SGPT) (U/L)- Day 364 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)- Day 14: number analyzed (Participants) | 5 | 10 | 2 | 20 | 18 | 20 | 20 | 9 | 10 | 10 | 2
  Creatinine (mg/dL)- Day 14 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)- Day 70: number analyzed (Participants) | 5 | 10 | 2 | 20 | 17 | 18 | 20 | 9 | 10 | 10 | 2
  Creatinine (mg/dL)- Day 70 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL)- Day 364: number analyzed (Participants) | 5 | 10 | 2 | 20 | 16 | 20 | 20 | 9 | 10 | 10 | 2
  Creatinine (mg/dL)- Day 364 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: The number (percentage) of Participants Reporting Unsolicited Adverse Events (AEs) was summarized by arm
Time Frame: Measured through Month 14 (Part A without second boost) or Month 18 (Part A with second boost, Part B, Part C)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part C, Group T7 | Part C, Group T8 | Part C, Group C3
Number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Participants
  Mild | 1 | 4 | 1 | 4 | 6 | 5 | 3 | 3 | 3 | 1 | 0
  Moderate | 2 | 3 | 0 | 11 | 8 | 9 | 11 | 4 | 6 | 5 | 1
  Severe | 1 | 1 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0
  Potentially life-threatening | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: The number (percentage) of participants with early discontinuation of vaccinations and reason for discontinuation was summarized by arm
Time Frame: Measured through Month 2 (Part A without second boost) or Month 6 (Part A with second boost, Part B, Part C)
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part C, Group T7 | Part C, Group T8 | Part C, Group C3
Number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Participants
  Withdrawal by Subject | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Investigator decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Participant refused study product administration | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Lost to Follow-Up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Unsolicited adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Participant unable to adhere to visit schedule | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Solicited adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Relocated, however participant agreed to continued follow-up with phone calls | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Did not discontinue SPA | 4 | 9 | 2 | 19 | 15 | 20 | 19 | 9 | 8 | 9 | 2

7. Primary Outcome: Number of Participants With Early Study Termination and Reason for Early Study Termination
Description: The number (percentage) of participants with early study termination and reason for early study termination was summarized by arm
Time Frame: Measured through Month 8 (Part A without second boost) or Month 12 (Part A with second boost, Part B, Part C)
Population: Started (enrolled).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part C, Group T7 | Part C, Group T8 | Part C, Group C3
Number analyzed (Participants) | 5 | 10 | 2 | 20 | 19 | 20 | 20 | 9 | 10 | 10 | 2
Participants
  Participant refused further participation | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Unable to contact participant | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Participant relocated, no follow-up planned | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Scheduled exit visit/end of study | 5 | 8 | 2 | 18 | 16 | 20 | 19 | 9 | 9 | 10 | 2

ADVERSE EVENTS:
Time Frame: The AE reporting period for this study comprises the entire study period for each individual participant (from the participant's study enrollment until his or her study completion or discontinuation), up to 18 months
Description: The number (percentage) of Participants Reporting Solicited AEs and unsolicited AEs including All-Cause Mortality, Serious Adverse Events (SAEs), and Other (Not Including Serious) Adverse Events were summarized by arm
Arm/Group | Part A, Group T1 | Part A, Group T2 | Part A, Group C1 | Part B, Group T3 | Part B, Group T4 | Part B, Group T5 | Part B, Group T6 | Part B, Group C2 | Part B, Group T7 | Part B, Group T8 | Part B, Group C3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10 | 0/2 | 0/20 | 0/19 | 0/20 | 0/20 | 0/9 | 0/10 | 0/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/10 | 0/2 | 1/20 | 0/19 | 1/20 | 0/20 | 0/9 | 0/10 | 0/10 | 0/2
Other Adverse Events (participants affected / at risk) | 5/5 | 10/10 | 1/2 | 19/20 | 19/19 | 20/20 | 20/20 | 9/9 | 10/10 | 10/10 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group T1 (N=5) | Part A, Group T2 (N=10) | Part A, Group C1 (N=2) | Part B, Group T3 (N=20) | Part B, Group T4 (N=19) | Part B, Group T5 (N=20) | Part B, Group T6 (N=20) | Part B, Group C2 (N=9) | Part B, Group T7 (N=10) | Part B, Group T8 (N=10) | Part B, Group C3 (N=2)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar artery dissection (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group T1 (N=5) | Part A, Group T2 (N=10) | Part A, Group C1 (N=2) | Part B, Group T3 (N=20) | Part B, Group T4 (N=19) | Part B, Group T5 (N=20) | Part B, Group T6 (N=20) | Part B, Group C2 (N=9) | Part B, Group T7 (N=10) | Part B, Group T8 (N=10) | Part B, Group C3 (N=2)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Solicited) (Gastrointestinal disorders) | 2 (2) | 7 (7) | 0 (0) | 3 (3) | 12 (12) | 4 (4) | 5 (5) | 0 (0) | 7 (7) | 8 (8) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (Solicited) (General disorders) | 3 (3) | 6 (6) | 0 (0) | 3 (3) | 16 (16) | 6 (6) | 1 (1) | 1 (1) | 10 (10) | 5 (5) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (Solicited) (General disorders) | 2 (2) | 3 (3) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Injection site pain (Solicited) (General disorders) | 5 (5) | 10 (10) | 1 (1) | 15 (15) | 19 (19) | 16 (16) | 19 (19) | 5 (5) | 10 (10) | 10 (10) | 0 (0)
Injection site swelling (Solicited) (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Injury associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (Solicited) (General disorders) | 5 (5) | 10 (10) | 0 (0) | 14 (14) | 18 (18) | 15 (15) | 13 (13) | 6 (6) | 9 (9) | 10 (10) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 7 (7) | 5 (5) | 8 (8) | 4 (5) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mycoplasma genitalium infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Solicited) (Investigations) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 16 (16) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Solicited) (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7) | 0 (0) | 0 (0) | 14 (14) | 3 (3) | 4 (4) | 0 (0) | 8 (8) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (9) | 0 (0) | 4 (4) | 17 (17) | 7 (7) | 5 (5) | 3 (3) | 9 (9) | 8 (8) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain fog (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Solicited) (Nervous system disorders) | 5 (5) | 10 (10) | 0 (0) | 10 (10) | 17 (17) | 8 (8) | 10 (10) | 4 (4) | 8 (8) | 9 (9) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spermatocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fixed eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT04177355/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT04177355/SAP_001.pdf